CLINICAL TRIAL: NCT06796647
Title: The Use of a Novel ESAT6/CFP10 Skin Test in Diagnosis of Latent Tuberculosis Infection Among Rheumatologic Patients
Brief Title: ESAT6/CFP10 Skin Testing for TB Infection in Rheumatologic Patients
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shui-Shan Lee, MD, Professor, Chinese University of Hong Kong
Other Study IDs: HMRF23220212
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis (TB)
Keywords: tuberculosis; skin testing; ESAT6/CFP10; rheumatology patients
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group: Adult patients with diagnosed rheumatologic diseases scheduled to receive b/tsDMARDs therapy
  Interventions: Diagnostic Test: ESAT6/CFP10 skin test

INTERVENTIONS:
Diagnostic Test: ESAT6/CFP10 skin test — Each recruited participant would be offered standard tuberculin skin test (TST) and ESAT6/CFP10 (C-TST) skin test on the same day or setting of clinical visit. TST and C-TST would be performed by the Mantoux technique with intradermal injection of 2U purified protein derivative-RT23 on one forearm and 5U (1.0µg/0.1 ml) of recombinant fusion protein ESAT6-CFP10 on the other forearm respectively.

SUMMARY:
The aim of the study is to pilot the application of a novel ESAT6/CFP10 (C-TST) skin test in rheumatologic disease patients prior to initiation of treatment with biologic and/or targeted synthetic disease-modifying antirheumatic drugs (b/tsDMARD). This is a prospective observational study involving the recruitment of patients with rheumatologic diseases who are planned for initiation of b/tsDMARD. Eligible patients would undergo skin testing by the Mantoux technique with purified protein derivative (PPD) RT23 on one forearm and C-TST on the other, alongside routine blood sampling for Interferon-Gamma Release Assay. The skin test results would be read within 48-72 hours afterwards. Treatment of TB infection would be provided in accordance with current clinical guidelines, followed by regular clinical monitoring for 2 years. Analyses involve performance evaluation of C-TST, and decision-analytical modelling incorporating multiple Markov process to evaluate the impact of management by LTBI testing methods on clinical outcomes and health care costs.

DETAILED DESCRIPTION:
Objective. The aim of the study is to pilot the application of a novel ESAT6/CFP10 (C-TST) skin test in rheumatologic disease patients prior to initiation of treatment with biologic and/or targeted synthetic disease-modifying antirheumatic drugs (b/tsDMARD), with the objectives of determining its performance and the cost-effectiveness of clinical management for latent tuberculosis infection (LTBI).

Design. A prospective observational study

Setting. Rheumatology Specialist clinic services in Hong Kong

Methods. This study involves the recruitment of patients with rheumatologic diseases who are planned for initiation of b/tsDMARD. Eligible patients would undergo skin testing by the Mantoux technique with intradermal injection of 2U purified protein derivative (PPD) RT23 on one forearm and 5U of C-TST on the other, alongside routine blood sampling for Interferon-Gamma Release Assay (IGRA) with QuantiFERON-TB Gold. The skin test results would be read within 48-72 hours afterwards. Treatment of LTBI would be provided in accordance with current clinical guidelines, followed by regular clinical monitoring for 2 years. Analyses involve performance evaluation of C-TST, and decision-analytical modelling incorporating multiple Markov process to evaluate the impact of management by LTBI testing methods on clinical outcomes and health care costs.

Main outcome measures. Concordance between different tests for LTBI by Kappa measure; sensitivity and specificity of C-TST test estimated with current standard; proportion of new TB cases averted, discounted QALYG and ICER.

Anticipated outcome. The study would provide preliminary evidence regarding the diagnostic performance of C-TST, and impact of its utilisation for treatment decision for rheumatologic diseases patients in the prevention of active tuberculosis diseases.

ELIGIBILITY:
Inclusion Criteria:

1. adult of age ≥ 18 and up to 65 years;
2. diagnosis of at least one classified rheumatologic disease; and
3. being planned to receive b/tsDMARDs therapy,
4. can communicate in Chinese and/or English.

Exclusion Criteria:

* diagnosis of active TB diseases,
* currently receiving TB or LTBI treatment;
* concurrent mental illnesses;
* prisoners.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatology patients followed up at the Specialist Services of regional hospitals in New Territories East Cluster in Hong Kong (Prince of Wales Hospital, Alice Ho Miu Ling Nethersole Hospital and North District Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
C-TST reading | from enrolment to reading test result at 48-72 hours
  Concordance between C-TST and standard TST
C-TST reading | from enrolment to reading test result at 2 weeks
  Concordance between C-TST and IGRA test result

SECONDARY OUTCOMES:
Proportion with TB disease | from enrolment to last followup at 2 years
  Proportion of patients by test results who developed TB disease

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, MD, Study Director — Chinese University of Hong Kong
Locations (2):
- S.H. Ho Research Centre for Infectious Diseases, Hong Kong, Hong Kong, China
- S.H. Ho Research Centre for Infectious Diseases, Shatin, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Access of individual level data at individual level is restricted for protection of privacy, as stipulated in the institutional approval